CLINICAL TRIAL: NCT00861302
Title: Evaluating Outcomes and Response Profiles of a Psychological Treatment for People With Chronic Pain
Brief Title: Evaluating a Chronic Pain Treatment Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSU094808B3E
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): This is the only group in the study. It consists of patients with chronic musculoskeletal pain who are receiving the treatment program
  Interventions: Behavioral: Mind-body emotional awareness program

INTERVENTIONS:
Behavioral: Mind-body emotional awareness program — This intervention, developed and offered by Dr. Howard Schubiner of St. John Providence Health System, consists of a single individual session with him, followed by four, classroom group sessions. The intervention includes expressive writing, mindfulness, and other techniques designed to enhance awareness and acceptance of the emotional factors underlying the chronic pain problem.

SUMMARY:
This interventional study seeks to evaluate the overall outcomes of a novel, emotional awareness intervention for people with chronic musculoskeletal pain and determine which patients benefit the most from this intervention. The investigators also are evaluating the effects of brief emotional communication technique embedded in the pre-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic musculoskeletal pain, not accounted for by disease or tissue pathology, who are seeking or referred for this psychological treatment program

Exclusion Criteria:

* Autoimmune diseases
* Cancer pain
* Illiterate
* Cognitively impaired
* Too medically ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | baseline, post-treatment, 3- and 6-month follow-ups

SECONDARY OUTCOMES:
Center for Epidemiologic Studies--Depression Scale | baseline, post-treatment, 3- and 6-month follow-ups
Satisfaction with Life Scale | baseline, post-treatment, 3- and 6-month follow-ups
McGill Pain Questionnaire | baseline, post-treatment, 3- and 6-month follow-ups
Impact of Events Scale-Revised | baseline, post-treatment, 3- and 6-month follow-ups
Positive Affect Negative Affect Scale-Expanded Version | baseline, post-treatment, 3- and 6-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Lumley, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- St. John Providence Health System, Southfield, Michigan, United States

REFERENCES:
- [Derived] Burger AJ, Lumley MA, Carty JN, Latsch DV, Thakur ER, Hyde-Nolan ME, Hijazi AM, Schubiner H. The effects of a novel psychological attribution and emotional awareness and expression therapy for chronic musculoskeletal pain: A preliminary, uncontrolled trial. J Psychosom Res. 2016 Feb;81:1-8. doi: 10.1016/j.jpsychores.2015.12.003. Epub 2015 Dec 11. PMID 26800632